CLINICAL TRIAL: NCT06289023
Title: Hippocampal Avoidance Whole Brain Irradiation With Simultaneous Integrated Boost for the Treatment of Lung Cancer Brain Metastases：A Prospective Phase II Study
Brief Title: HA-WBRT-SIB for Brain Metastasis of Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, ZONG MEI ZHOU, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC1278
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Lung Neoplasm; Brain Metastases; Simultaneous Integrated Boost; Hippocampal Avoidance; Cognitive Function
Keywords: Lung Neoplasm; Brain Metastases; Simultaneous integrated boost; Hippocampal avoidance; Cognitive function
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HA-WBRT-SIB (Experimental): Patients with lung cancer and brain metastases undergo HA-WBRT-SIB using image-guided radiotherapy, receiving a total dose of 30-36 Gy delivered in 18-20 fractions to the whole brain (CTV), while the dose to the GTV is boosted to 44 Gy-52 Gy in 18-20 fractions, ﬁve times a week. The optimal mean dose (Dmean) to the bilateral hippocampus should optimally be ≤ 8 Gy, with a mandatory maximum dose (Dmax) to the hippocampus not exceeding 10 Gy; the preferred Dmean to the hippocampus PRV should optimally be ≤ 9 Gy, while the mandatory Dmax to the hippocampus PRV should be ≤ 12 Gy. The HVLT-R immediate recall scores are obtained at baseline and 1, 3, and 6 months after treatment.
  Interventions: Radiation: HA-WBRT-SIB

INTERVENTIONS:
Radiation: HA-WBRT-SIB — A total dose of 30-36 Gy delivered in 18-20 fractions to the whole brain (CTV), while the dose to the GTV were boosted to 44 Gy-52 Gy in 18-20 fractions, ﬁve times a week.

SUMMARY:
Patients with lung cancer and brain metastases undergo HA-WBRT-SIB using image-guided radiotherapy, receiving a total dose of 30-36 Gy delivered in 18-20 fractions to the whole brain (CTV), while the dose to the GTV is boosted to 44 Gy-52 Gy in 18-20 fractions, ﬁve times a week. The optimal mean dose (Dmean) to the bilateral hippocampus should optimally be ≤ 8 Gy, with a mandatory maximum dose (Dmax) to the hippocampus not exceeding 10 Gy; the preferred Dmean to the hippocampus PRV should optimally be ≤ 9 Gy, while the mandatory Dmax to the hippocampus PRV should be ≤ 12 Gy. The HVLT-R immediate recall scores are obtained at baseline and 1, 3, and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically diagnosed primary lung cancer with brain metastasis confirmed via magnetic resonance imaging (MRI);
2. 18-75 years old;
3. BM outside a 10 mm margin around either hippocampus;
4. at least one BM existed if prior resection of BM was done;
5. BM measuring less than 5.0 cm in maximal extent;
6. Eastern Cooperative Oncology Group (ECOG) performance status scores of 0-2

Exclusion Criteria:

1. previous brain radiotherapy or brain metastasis resection;
2. history of malignancies other than lung cancer;
3. radiographic evidence of hydrocephalus or other architectural distortion of the ventricular system, leptomeningeal metastases
4. presence of other serious illnesses such as acute myocardial infarction, severe arrhythmia, or psychiatric disorders within the past 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
OS | 24 months
  the time from the end of brain radiotherapy to death from any cause

SECONDARY OUTCOMES:
PFS | 24 months
  the time from the end of brain radiotherapy to tumor progression or death from any cause
iPFS | 24 months
  the time from the end of brain radiotherapy to intracranial tumor progression or death from any cause
HVLT-R learning score | at baseline and 1, 3, and 6 months after radiotherapy
  The HVLT scores were calculated as the sum of trials 1, 2, and 3

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciecnces and Peking Union Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li Z, Wang J, Deng L, Zhai Y, Zhang T, Bi N, Wang J, Wang X, Liu W, Xiao Z, Chen D, Lv J, Feng Q, Wang W, Zhou Z. Hippocampal avoidance whole-brain radiotherapy with simultaneous integrated boost in lung cancer brain metastases and utility of the Hopkins verbal learning test for testing cognitive impairment in Chinese patients: a prospective phase II study. BMC Cancer. 2024 Jul 26;24(1):899. doi: 10.1186/s12885-024-12559-1. PMID 39060968